CLINICAL TRIAL: NCT02895672
Title: A Real-world, Observational Study of GLP-1 Therapy Added to Basal Insulin in Patients With Type 2 Diabetes Mellitus
Brief Title: GLP-1/Basal Insulin Combination Therapy
Status: Completed | Type: Observational
Sponsor: Albany College of Pharmacy and Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 15-026
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weekly GLP-1 therapy: exenatide: Patients receiving weekly exenatide
  Interventions: Drug: GLP-1 therapy
- Daily GLP-1 therapy liraglutide: Patients receiving daily liraglutide
  Interventions: Drug: GLP-1 therapy

INTERVENTIONS:
Drug: GLP-1 therapy — The investigators will assess the efficacy and safety of 12 months of GLP-1 therapy added to the therapeutic regimen of a group of T2DM patients who have received basal insulin therapy for a minimum of one year.
  Other Names: Bydureon, Victoza

SUMMARY:
This is a real-world, pre-post observational study from an ambulatory endocrinology practice which will determine the effectiveness and safety of the addition of glucagon-like peptide-1(GLP-1) agonist therapy (weekly exenatide {Bydureon} or daily liraglutide {Victoza}), added to the regimens of T2DM patients who have already received a minimum of one year of basal insulin therapy. Specifically, the investigators hypothesize that GLP-1 agonist therapy added to basal insulin therapy will result in statistically significant improved glycemic control and weight loss, with no higher risk of hypoglycemia compared to baseline.

DETAILED DESCRIPTION:
This is a pre-post observational study which will assess the efficacy and safety of 12 months of GLP-1 therapy added to the therapeutic regimen of a group of T2DM patients. This study was reviewed and approved by the Albany College of Pharmacy and Health Sciences Institutional Review Board. Potential subjects will be identified via a computerized text search of the medication and problem fields of patient electronic medical records (EMR). Search terms include exenatide, Bydureon, liraglutide, Victoza, GLP-1 agonist, NPH, Lantus, Levemir, and T2DM. Individual records of identified patients will be reviewed to ascertain if all applicable study criteria are met. Inclusion criteria are: T2DM, age 18-85 years, documentation of basal insulin therapy for minimum of one year prior to GLP-1 initiation, and addition of weekly exenatide or daily liraglutide added to basal insulin therapy for a minimum of 12 months. Exclusion criteria include: Type 1 diabetes, patients receiving prescription medications for weight loss, and initiation of additional diabetes, hypertension or cholesterol drugs during the follow-up period.

A data collection form will be utilized to collect the following patient information: baseline demographic information (gender, age, height, weight), duration of diabetes, medications, laboratory information (HbA1C, cholesterol profile [total cholesterol, triglycerides, LDL-C, HDL-C]), and blood pressure. The primary study outcome is change in HbA1C from baseline to 12 months after GLP-1 therapy is added to basal insulin therapy. A separate analysis including patients who do not complete 12 months of GLP-1 therapy will also be performed. Secondary outcomes are change in weight, percentage of patients achieving an A1C of <7%, changes in systolic and diastolic blood pressures, changes in lipid parameters (TC, LDL-C, HDL-C, and TG's), and reductions in number/doses of diabetes, blood pressure, and lipid lowering medications. Safety will be assessed by collection of reported adverse effects. Medication compliance will be assessed by review of an insurance data base record of refills.

ELIGIBILITY:
Inclusion Criteria:

* T2DM, age 18-85 years, documentation of basal insulin therapy for minimum of one year prior to GLP-1 initiation, and addition of weekly exenatide or daily liraglutide added to basal insulin therapy

Exclusion Criteria:

* Type 1 diabetes, patients receiving prescription medications for weight loss, and initiation of additional diabetes, hypertension or cholesterol drugs during the follow-up period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pre-post observational study which will assess the efficacy and safety of 12 months of GLP-1 therapy added to the therapeutic regimen of a group of T2DM patients from a community endocrinology practice who have received basal insulin therapy for a minimum of one year.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
A1C | 12 months
  from baseline to 12 months after GLP-1 therapy is added to basal insulin therapy

IPD SHARING:
Plan to Share IPD: Undecided